CLINICAL TRIAL: NCT01794026
Title: Use of Diffusion Weighted Magnetic Resonance Imaging to Stage Gastric Adenocarcinoma Patients Preoperatively
Brief Title: Diffusion Weighted Magnetic Resonance Imaging for Preoperative Staging in Gastric Adenocarcinoma Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DWMRIGASTADENO
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2013-12

CONDITIONS: Gastric Adenocarcinoma
Keywords: diffusion weighted; magnetic resonance imaging; surgery; histopathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diffusion MRI (Experimental): histopathology of lymph nodes diagnosed by diffusion weighted magnetic resonance imaging
  Interventions: Procedure: diffusion weighted magnetic resonance imaging

INTERVENTIONS:
Procedure: diffusion weighted magnetic resonance imaging — for diagnostic purposes, diffusion weighted magnetic resonance imaging in all patients

SUMMARY:
Preoperative staging for gastric adenocarcinoma is an important procedure to detect advanced disease stateS for the patients in which the surgery may be unnecessary to perform. Although there are many imaging techniques for this purpose, sensitivity and specificity of these techniques still remains to be low.Preoperative detection of peritoneal carcinomatosis and involvement of lymph nodes beyond D2 may prevent surgical procedures.

Removal of the determined lymph nodes according to the type of the surgery is the accepted surgical method. However, accurate determination of malignant lymph nodes may prevent dissection of some groups of the lymph nodes. These findings may cause a new definition of gastric lymph node dissection.

DETAILED DESCRIPTION:
1. proven endoscopic diagnosis of gastric adenocarcinoma
2. for staging purposes, computed tomography for all patients
3. evaluation of benign and malignant lymph nodes according to computed tomography findings and mapping of the lymph nodes
4. to state precisely resectable patients according to computed tomography and anesthetic evaluation
5. evaluation of benign and malignant lymph nodes according to diffusion weighted magnetic resonance imaging findings and mapping of the lymph nodes
6. standard gastrectomy and D2 lymph node dissection
7. mapping of the lymph nodes after taking the specimen out
8. histopathological diagnosis of the lymph nodes and mapping
9. comparison of the results taken from computed tomography, diffusion weighted magnetic resonance imaging and histopathological analysis

ELIGIBILITY:
Inclusion Criteria:

* gastric adenocarcinoma proven by endoscopic biopsy;
* application of both computed tomography and diffusion weighted magnetic resonance imaging;
* standard gastrectomy and a D2 lymph node dissection;
* desire to attend the study protocol

Exclusion Criteria:

* preoperative neoadjuvant therapy;
* metastatic disease;
* undesired reaction to attend the study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
efficacy of diffusion weighted magnetic resonance imaging to detect benign and malignant lymph nodes | one year
  to compare the radiologic diagnosis of benign and malignant lymph nodes with histopathological diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University Faculty of Medicine Dept of General Surgery, Istanbul, Turkey (Türkiye)